CLINICAL TRIAL: NCT04122118
Title: Pharmacist-led Transitions of Care in the Outpatient Oncology Infusion Center
Brief Title: Pharmacist-led Transitions of Care in the Outpatient Oncology Infusion Center for Patients With Solid Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19D.411; JT 13521 (Other: JeffTrial Number)
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hearth services research (pharmacist-led education) (Experimental): PHASE I: Patients' medical records are reviewed.
  PHASE II: Patients receive pharmacist-led education on antineoplastic therapies including what to expect during infusion, general drug facts, common adverse effects, side effect management, and when to contact provider.
  Interventions: Other: Medical Chart Review; Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review
Other: Educational Intervention — Receive pharmacist-led education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Educational
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies how well pharmacist-led transitions of care works in the outpatient oncology infusion center for patients with solid tumor. Having a pharmacist in the outpatient oncology infusion center may help to identify and correct medical related problems and improve overall patient and staff satisfaction. Patients receiving education may benefit from gaining a better understanding of their antineoplastic therapy. Understanding the side effects associated with the therapy may also help patients better be prepared to manage any adverse effects they may experience.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate the effectiveness of a clinical oncology pharmacist in the outpatient infusion center through education, and the identification and correction of medication related problem (MRP)s.

SECONDARY OBJECTIVE:

I. To evaluate overall patient and staff satisfaction with the added clinical oncology pharmacy education.

EXPLORATORY OBJECTIVE:

I. Estimate the cost avoidance utilizing the pharmacy services provided in the prospective trial.

OUTLINE:

PHASE I: Patients' medical records are reviewed.

PHASE II: Patients receive pharmacist-led education on antineoplastic therapies including what to expect during infusion, general drug facts, common adverse effects, side effect management, and when to contact provider.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor diagnosis
* Starting day 1 of new antineoplastic infusion
* English speaking (and/or English-speaking primary caregiver/proxy)

Exclusion Criteria:

* Metastasis to the brain and/or central nervous system (CNS) with evidence of impaired cognition
* Severe cognitive impairment including dementia with inability to consent to the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Number of medical related problem (MRP)s identified by the pharmacist through retrospective chart reviews (Phase I) | Up to 1 year
  MRPs will be assigned to a specific category and the total number of MRPs in each category will be recorded. Categories include but are not limited to: incorrect dose, therapeutic duplication, drug not indicated, drug interaction, monitoring recommendation, drug allergy, or potential for adverse event.
Percent of MRPs corrected as a result of the clinical oncology pharmacist services (Phase II) | Up to 1 year
  In phase 2 (prospective) MRPs will also be recorded and categorized, but in addition the outcomes relating to each MRP pharmacist intervention will be recorded. MRPs found by the pharmacist will be communicated to the patient's oncologist or primary care provider, and the pharmacist will follow-up to see if changes were made.

SECONDARY OUTCOMES:
Patient and provider satisfaction with the pharmacist-led education | Up to 1 year
  The survey results will help determine the need for a clinical oncology pharmacist in the outpatient infusion center. Satisfaction will be assessed using a Likert-scale survey. Scale ranges from 1 (strongly disagree) to 5 (strongly agree).

OTHER OUTCOMES:
Estimate of Cost avoidance utilizing pharmacy services | Up to 1 year
  In order to determine cost avoidance the type of interventions made and the time associated with each intervention will be recorded. The cost per intervention will be calculated by multiplying the pharmacist salary in minutes by the time for each intervention. The intervention types will be assigned cost avoidance values based on previous literature and these will be used to determine the cost benefit for the interventions made during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Espinosa, PharmD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No